CLINICAL TRIAL: NCT01900210
Title: Sustainable Disease Risk Reduction Strategies for CJ Systems
Brief Title: Sustainable HIV Risk Reduction Strategies for CJ Systems
Acronym: DRR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne Lehman (Other)
Responsible Party: Sponsor-Investigator, Wayne Lehman, Senior Research Scientist, Texas Christian University
Organization: Texas Christian University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA25885-Sum08-13
Record Dates: First submitted 2013-07-02; First posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: HIV Risk Behaviors
Keywords: Criminal justice; substance abuse treatment; HIV risk behaviors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- WaySafe (Experimental): WaySafe -- Participants in this arm received a curriculum titled WaySafe that focused on identifying, planning for, and avoiding HIV risk behaviors after release from prison. WaySafe included 6 hour-long, group-based, highly interactive sessions normally held weekly with homework assignments given between sessions.
  Interventions: Behavioral: WaySafe
- Treatment as usual (No Intervention): Participants in this arm completed pre- and post-surveys and attended normal substance abuse programming.

INTERVENTIONS:
Behavioral: WaySafe
  Arms: WaySafe

SUMMARY:
The purpose of the Texas Christian University (TCU) Disease Risk Reduction (DRR) Project is to develop and test an intervention designed to increase positive decision-making skills among offenders for healthy living, including skills for making decisions for reducing disease risk behaviors, particularly those involving HIV and Hepatitis B & C. This project focuses on the critical transition time between incarceration and return to the community.

DETAILED DESCRIPTION:
The purpose of the TCU DRR Project is to develop and test an intervention designed to increase positive decision-making skills among offenders for healthy living, including skills for making decisions for reducing disease risk behaviors. This project focuses on risky sexual and drug use behaviors during re-entry, including problem recognition, commitment to change, and strategies for avoiding behavioral risks of infections. Motivational and planning sessions will be delivered near the end of criminal justice (CJ) institution-based substance abuse treatment, and they will also bridge into re-entry care services during community transitional treatment by using a self-study toolkit for released offenders that emphasize applications of DRR principles. This 5-year project has been funded by the National Institute on Drug Abuse.

The intervention has two components - an in-prison and a post-release component.

• The in-prison component, WaySafe, is a six session, manual-based training on decision-making skills that occurs during the last several months of treatment before release from incarceration. It is a group-based, interactive curriculum based on TCU Mapping Enhanced Counseling strategies, which are used to visually enhance communication between clients and counselors. Homework assignments are given to be completed between the weekly sessions. The six hour-long WaySafe sessions are conducted by current counselors at the facility who have been trained in the curriculum.

For comparison purposes, some offenders who voluntarily agree to participate in the DRR study are randomly assigned to attend "treatment as usual." All participants in the study first sign an Informed Consent document indicating that their participation is voluntary and that they have been informed about their rights as research participants. They are also asked to complete a brief pre-test at the beginning of the study and a brief post-test at the end of the six-week period. A signed Certificate of Completion is given to all participants who complete the study.

• The post-release component, Keep It Safe, is a self-study toolkit given to offenders when they are released from incarceration, using mapping principles similar to those in the WaySafe sessions. It is designed to reinforce decision-making skills during this transition period and includes multiple assignments on topics such as risk taking, making better decisions regarding risky behaviors, and decisions regarding HIV testing.

For comparison purposes, some offenders are randomly selected to receive a booklet that includes readings on HIV and Hepatitis B&C derived from National Institutes of Health (NIH) and Center for Disease Control (CDC) materials, with short quizzes after each section. Both the Keep It Safe and CDC Readings booklets are designed to take about five hours to complete including a final follow-up survey in each booklet. Offenders are asked to mail their completed booklets directly to TCU in a provided pre-addressed, franked envelope. A Certificate of Completion is mailed directly to the participant when the completed workbook and follow-up survey is received at TCU project offices.

ELIGIBILITY:
Inclusion Criteria:

* Incarcerated offenders in eight participating facilities in two states entering the last phase of their prison-based substance abuse treatment.

Exclusion Criteria:

* Sex offenders or those convicted of a violent crime.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1396 (Actual)
Dates: Start 2008-08; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
HIV Knowledge Confidence (change from pre-test to post-test) | One week prior to the intervention start (for both experiemental and control arms) and one week after the intervention
  13 item scale comprised of items assessing knowledge, confidence and motivation regarding HIV knowledge (alpha = .89. Responses on a 5-point "strongly disagree" to "strongly agree" scale. Sample item -- "You should know enough to teach others what they should do if they have been exposed to HIV."
Avoiding Risky Sex (change from pre-test to post-test) | One week prior to the intervention start (for both experiemental and control arms) and one week after the intervention
  13 item scale comprised of items assessing knowledge, confidence and motivation regarding avoiding risky sex behaviors (alpha = .91. Responses on a 5-point "strongly disagree" to "strongly agree" scale. Sample item -- "You have learned to think ahead in order to make less risky decisions about sex."
Avoiding Risky Drug Use (change from pre-test to post-test) | One week prior to the intervention start (for both experiemental and control arms) and one week after the intervention
  12 item scale comprised of items assessing knowledge, confidence and motivation regarding avoiding risky drug use behaviors (alpha = .85. Responses on a 5-point "strongly disagree" to "strongly agree" scale. Sample item -- "If you decide to inject drugs, you will always use a 'clean needle'."
HIV Testing Awareness (change from pre-test to post-test) | One week prior to the intervention start (for both experiemental and control arms) and one week after the intervention
  7 item scale comprised of items assessing knowledge and motivation regarding getting tested for HIV (alpha = .76). Responses on a 5-point "strongly disagree" to "strongly agree" scale. Sample item -- "You plan on being tested regularly for HIV."
Risk Reduction Skills (change from pre-test to post-test) | One week prior to the intervention start (for both experiemental and control arms) and one week after the intervention
  14 item scale comprised of items assessing knowledge, confidence and motivation regarding identifying, planning for, and avoiding risk situations (alpha = .85). Responses on a 5-point "strongly disagree" to "strongly agree" scale. Sample item -- "You know how to stand up for yourself when pressured to take a risk."

CONTACTS AND LOCATIONS:
Overall Officials: Wayne E Lehman, Ph.D., Principal Investigator — Institute of Behavioral Research, Texas Christian University